CLINICAL TRIAL: NCT01233505
Title: A Phase I Study of ABT-888 in Combination With Oxaliplatin and Capecitabine in Advanced Solid Tumors
Brief Title: Veliparib, Oxaliplatin, and Capecitabine in Treating Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02543; NCI-2011-02543 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000687938; C010903 (Other: University of Wisconsin Hospital and Clinics); 8604 (Other: CTEP); P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2013-10

CONDITIONS: Adenocarcinoma of the Pancreas; Adenocarcinoma of the Stomach; BRCA1 Mutation Carrier; BRCA2 Mutation Carrier; Ovarian Mucinous Cystadenocarcinoma; Recurrent Breast Cancer; Recurrent Colon Cancer; Recurrent Gastric Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Pancreatic Cancer; Recurrent Rectal Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Gastric Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Pancreatic Cancer; Stage IV Rectal Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Rectal Neoplasms | interventions — veliparib; Capecitabine; Oxaliplatin

ARMS (1):
- Treatment (veliparib, capecitabine, oxaliplatin) (Experimental): Patients receive veliparib PO twice daily and capecitabine PO twice daily on 1-7 and 15-21, and oxaliplatin IV over 2 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: veliparib; Drug: capecitabine; Drug: oxaliplatin; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: veliparib — Given PO
  Other Names: ABT-888
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and the best dose of veliparib when given together with capecitabine and oxaliplatin in treating patients with advanced solid tumors. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving veliparib together with capecitabine and oxaliplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicities (DLTs) and the maximum tolerated dose (MTD) of ABT-888 (veliparib) in combination with oxaliplatin and capecitabine in advanced solid tumors.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of ABT-888, oxaliplatin, and capecitabine when administered concomitantly.

II. To evaluate the safety and tolerability of the ABT-888 in combination with capecitabine and oxaliplatin.

III. To assess for evidence of anti-tumor activity with this combination, per tumor measurements using RECIST criteria, in these patients.

TERTIARY OBJECTIVES:

I. To assess the inhibition of poly(ADP-ribose) polymerase (PARP) in peripheral blood mononuclear cells secondary to treatment with ABT-888.

II. To determine the pharmacokinetics of ABT-888 in combination with oxaliplatin and capecitabine and the relation to treatment side effects.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive veliparib orally (PO) twice daily and capecitabine PO twice daily on 1-7 and 15-21, and oxaliplatin intravenously (IV) over 2 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and urine sample collection at baseline and periodically during study for pharmacokinetic and poly (ADP-ribose) polymerase (PARP) inhibition studies.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumors that fulfill ≥ 1 of the following criteria:

  * BRCA1/2 mutation and a BRCA-related malignancy

    * Patients without a known BRCA mutation must have a probability of harboring a BRCA gene mutation as assessed by BRCAPRO computer program
    * Patients with a probability of having genetic mutation ≥ 20% or a BRCA mutation based on a non-Myriad test, must have a formal BRCA testing by Myriad Genetic Laboratories
    * Patients with known deleterious BRCA 1 or 2 mutation or a mutation of uncertain significance
    * Patients who refuse BRCA testing not allowed unless they have another acceptable histology
  * First- or second-line metastatic colorectal cancer
  * Any-line metastatic mucinous ovarian cancer
  * Any line of other metastatic gastrointestinal malignancies in which oxaliplatin has shown some activity (i.e., gastric or pancreatic adenocarcinoma)
* Patients with uncontrolled CNS metastasis are not eligible; patients with CNS metastases who have had them treated and are stable for > 3 months will be eligible; patients must be off steroid treatment prior to study enrollment
* Measurable disease

  * Patients with ovarian cancer who have a pre-treatment CA 125 level of at least twice the upper limit of normal allowed
* ECOG performance status (PS) 0-2 (Karnofsky 60-100%)
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver metastases)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Fertile patients must use adequate contraception (i.e., hormonal, barrier method of birth control, or abstinence)
* Not pregnant or nursing
* Negative pregnancy test
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib or other agents used in study
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No history of positive serology for hepatitis A, B, or C, liver disease, or other forms of hepatitis or cirrhosis
* Patients who have active seizures or history of seizures are ineligible
* No condition that impairs the ability to swallow and retain veliparib capsules, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction
* No peripheral neuropathy ≥ grade 2
* No prolonged QTC > 450 msec (male) or QTC > 470 (female)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Recovered from adverse events of prior therapy or prior surgical procedures

  * Patients with chronic grade 1 or 2 adverse events that are not expected to improve are allowed at investigator's discretion
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 4 weeks since prior radiotherapy with no > 35% of marrow irradiation
* Prior fluoropyrimidine allowed
* Prior veliparib allowed provided it was part of a single- or limited-dosing study, such as a phase 0 study
* Prior capecitabine allowed provided patient tolerated 3500 mg/m² for 7 days out of 14 days
* No other prior investigational agents
* No prior oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated (MTD) dose of veliparib in combination with oxaliplatin and capecitabine as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days
  MTD defined as the dose level at which less than one-third of patients experience a dose-limiting toxicity (DLT).
Dose-limiting toxicities of veliparib in combination with oxaliplatin and capecitabine as assessed by NCI CTCAE version 4.0 | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics of veliparib administered concomitantly with oxaliplatin and capecitabine | At baseline, at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours of days 1 and 7
  Graphical displays of individual, mean, and median plasma concentration over time will be presented at each ABT-888 dose level and overall in the entire group. Descriptive summaries for each pharmacokinetic endpoint will be presented by ABT-888 dose level.
Safety and tolerability as assessed by NCI CTCAE version 4.0 | Up to 30 days
  Reported in tabular format, both per dose level, as well as in the aggregate cohort.
Anti-tumor response according to Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 30 days
  Anti-tumor responses will be summarized using descriptive statistics and will be presented in tables. In addition, two-sided 90% confidence intervals for the proportions of subjects with a confirmed anti-tumor response will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States